CLINICAL TRIAL: NCT00455754
Title: Double-Blind, Randomized, Placebo-Controlled Multicenter Trial on the Efficacy of Esomeprazole Treatment for Patients With Lymphocytic Gastritis
Brief Title: Esomeprazole Treatment for Patients With Lymphocytic Gastritis
Acronym: LYNEX
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Technische Universität Dresden (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LYNEX
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-02

CONDITIONS: Lymphocytic Gastritis
MeSH Terms: interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Esomeprazole

SUMMARY:
The purpose of this study is to determine whether treatment with esomeprazole alone is able to heal patients with lymphocytic gastritis

DETAILED DESCRIPTION:
Recently, a placebo controlled trial of our group has shown that H. pylori eradication therapy consisting of omeprazole 20 mg bid, clarithromycin 500 mg bid, amoxicillin 1000 mg bid for seven days leads to a complete long-lasting resolution of lymphocytic gastritis in 96 % of patients. However, after 3 months we also found a healing rate of 50 % in patients who received omeprazole 20 mg bid and placebo antibiotics for seven days suggesting spontaneous remission or a potential PPI effect. Thus, we speculate that PPI therapy may have led to elimination of H. pylori and subsequently healing of lymphocytic gastritis in those patients with potentially minimal H. pylori colonization at baseline. For this reason we investigate whether a PPI treatment alone is able to heal patients with lymphocytic gastritis.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven lymphocytic gastritis (IEL > 25/100)
* Male or female aged 18 years or older
* Signed and written informed consent

Exclusion Criteria:

* Regular NSAID or aspirin intake
* Concomitant medication with antibiotics, bismuth subsalicylate, aminosalicylates
* Regular PPI therapy
* Treatment with ketoconazole or other CYP3A inhibitors
* previous surgery of the stomach
* known or suspected hypersensitivity to esomeprazole
* Malignant diseases
* Concomitant severe diseases
* Pregnancy or lactation
* Contraindication to take biopsies (Quick < 50%, PTT > 50 s, thrombocytes < 100.000/mm3)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2007-02; Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The primary objective is to assess the healing rate of
patients with lymphocytic gastritis irrespective of H. pylori status after treatment
with esomeprazole 20 mg twice daily for 2 weeks.

SECONDARY OUTCOMES:
Secondary objective of the study are to evaluate the grade and activity of gastritis before and after
treatment according to updated Sydney classification, to assess the clinical GI symptoms at baseline and after 3 months
and to evaluate influence of the H. pylori-Status

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Madisch, MD, Principal Investigator — Medical Department I, University Hospital Carl Gustav Carus, Technical University Dresden, Germany
Locations (1):
- Medical Department I, University Hospital Carl Gustav Carus, Technical University, Dresden, Germany